CLINICAL TRIAL: NCT03813810
Title: The Impact of Air Pollution on Chronic Respiratory Diseases: a Prospective Cohort Study
Brief Title: Impact of Air Pollution on Chronic Respiratory Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); SMG-SNU Boramae Medical Center (Other); National Medical Center, Seoul (Other); KangWon National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Air_pollution_cohort
Record Dates: First submitted 2018-12-23; First posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2018-12

CONDITIONS: Chronic Obstructive Pulmonary Disease; Asthma; Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, induced sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Normal: People without any chronic pulmonary diseases.
  Interventions: Other: Non
- Chronic obstructive pulmonary disease: Patients with chronic obstructive pulmonary disease.
  Interventions: Other: Non
- Asthma: Patients with asthma
  Interventions: Other: Non
- Idiopathic pulmonary fibrosis: Patients with idiopathic pulmonary fibrosis
  Interventions: Other: Non

INTERVENTIONS:
Other: Non — There would be no interventions. Only measurements will be performed.

SUMMARY:
The aim of this study is to evaluate the impact of air pollution on the occurrence and clinical course of chronic respiratory diseases, and discover new biomarkers from various devices such as CT images that can indicate the process and amount of lung damage caused by air pollution.

Accordingly, the investigators have designed an prospective cohort with enrollment of normal people and patients with chronic respiratory diseases of three different categories (chronic obstructive pulmonary disease, asthma, idiopathic pulmonary fibrosis). Participants will be followed up for a period of one year, with evaluation of the clinical course of the respiratory disease and exposure to air pollution.

DETAILED DESCRIPTION:
Normal people (n=90) and patients with chronic respiratory diseases (chronic obstructive pulmonary disease, asthma, idiopathic pulmonary fibrosis, n=90 for each disease) will be enrolled at 5 different institutions in South Korea and followed up for one year. Inspiratory-expiratory CTs and tests including physical examination and blood/urine tests would be performed at the time of enrollment and the time at completion of the follow up period for each participant. Participants would be checked for the residency and working places, as well as checked for the amount of air pollution exposure using a wearable measurement device for 5 days during the study period ( time at enrollment / 3 months / 6 months / 9 months / time at completion). The device would cause no effect on usual daily life or the medical status of the participant. The clinical course such as occurrence of disease, acute exacerbation, decline of lung function, imaging status, mortality would be evaluated as well as the exposure of air pollution for each individual.

ELIGIBILITY:
Inclusion Criteria:

* Normal: People with no lung lesions in chest X-ray and St. George's Respiratory Questionnaire score <25, and post bronchodilator FEV1/FVC (forced expiratory volume at one second/forced vital capacity) >= 0.7 and FEV1 >= 80% and FVC >= 80%.
* Chronic obstructive pulmonary disease: Patients with over 10 pack-years of smoking history and post bronchodilator FEV1/FVC <0.7 and FEV1 < 80%, and no other reason for decline of lung function.
* Asthma: Patients with FEV1/FVC < 0.85 and increase in over 12% and 200mL of FEV1 by bronchodilator inhalation. Patients with P20 < 16mg/dL by bronchial provocation test.
* Idiopathic pulmonary fibrosis: Shows usual interstitial pneumonia according to chest CT and has no other reasons such as systematic diseases or medication history.

Exclusion Criteria:

* Subjects who refused for enrollment in the study
* Subjects who experienced an acute exacerbation within 1 month.
* Subjects under age of 19.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal adults and adult patients with chronic respiratory disease (chronic obstructive pulmonary disease, asthma, idiopathic pulmonary fibrosis)
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2019-01-25 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Rate of mortality | an average of 1 year
  Events of mortality through study completion
Rate of acute exacerbations | an average of 1 year
  Events of acute exacerbations through study completion
Change of disease extent in CT imaging | an average of 1 year
  Emphysema index (0-100, higher values representing worse outcome)
Change in lung function | an average of 1 year
  FEV1 (forced expiratory volume at one second, 10-150 %, lower values representing worse outcome)
Change in symptom scor | an average of 1 year
  St. George's Respiratory Questionnaire score (0-100, higher values representing worse outcome)

IPD SHARING:
Plan to Share IPD: Undecided